CLINICAL TRIAL: NCT05302388
Title: A Phase I Randomized, Double-blind, Placebo-controlled, Dose-increasing Single Dose Study Evaluating the Safety, Tolerability，Pharmacokinetics and Pharmacodynamics Analysis of Pegloticase in Subjects With Asymptomatic Hyperuricemia
Brief Title: A Study Exploring Efficacy of Pegloticase in Subjects With Asymptomatic Hyperuricemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIBP-R002
Record Dates: First submitted 2022-03-19; First posted 2022-03-31 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Asymptomatic Hyperuricemia
Keywords: Hyperuricemia; Pegloticase; Safety; Tolerability
MeSH Terms: conditions — Hyperuricemia | interventions — Dexamethasone; Diphenhydramine

STUDY DESIGN:
Intervention Model Description: This is a phase I randomized, double-blind, placebo-controlled and dose-increasing single dosing study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the study period, the subjects and all personnel involved in the evaluation and analysis of the results were unaware of the actual grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Drug: SIBP-R002 & Dexamethasone/Methyl prednisolone & Diphenhydramine Starting from the lowest dose, when the former dose does not meet the termination criteria, then start the next dose group study until Maximum Tolerated Dose (MTD).
  Interventions: Drug: SIBP-R002; Drug: Dexamethasone or Methyl prednisolone; Drug: Diphenhydramine
- Placebo control group (Placebo Comparator): Placebo control: The same volume of placebo as SIBP-R002 & Dexamethasone/Methyl prednisolone & Diphenhydramine The rule and dose of placebo were the same as SIBP-R002.
  Interventions: Drug: Dexamethasone or Methyl prednisolone; Drug: Diphenhydramine; Drug: Placebo

INTERVENTIONS:
Drug: SIBP-R002 — SIBP-R002: injection; strength: 1, 2, 4, 8 or 12 mg; dose escalation and the first group is 1mg (intravenous infusion, 5 groups, the first group consisted of four people, and the other groups consisted of eight).
  Arms: Experimental group
Drug: Dexamethasone or Methyl prednisolone — Intravenous infusion, 5mg or 1~2mg/kg. These were administered within 30 minutes prior to infusion of the experimental drug.
Drug: Diphenhydramine — 10mg, intramuscular injection.These were administered within 30 minutes prior to infusion of the experimental drug.
Drug: Placebo — The same volume of placebo as SIBP-R002: injection; strength: the same volume of placebo as SIBP-R002 of 1, 2, 4, 8 or 12 mg (intravenous infusion, 5 groups, the first group consisted of one people, and the other groups consisted of two). The rule and dose of placebo were the same as SIBP-R002.
  Arms: Placebo control group

SUMMARY:
The main purpose To evaluate the safety and tolerability of pegloticase in subjects with asymptomatic hyperuricemia by single intravenous infusion at different doses, and to provide a basis for multiple doses of Pegloticase in subjects with asymptomatic hyperuricemia.

A secondary purpose To evaluate the pharmacokinetics, pharmacodynamics and immunogenicity of Pegloticase with single-pass intravenous drip in subjects with asymptomatic hyperuricemia.

Exploratory purpose Plasma uricase activity (pUox) analysis of pegloticase with single-pass intravenous drip in subjects with asymptomatic hyperuricemia.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics analysis of pegloticase in subjects with asymptomatic hyperuricemia.

This is a phase I randomized, double-blind, placebo-controlled and dose-increasing single dosing study. Five dose groups of 1, 2, 4, 8 or 12 mg were planned to explore the most appropriate dose and to provide a basis for multiple doses of Pegloticase in subjects with asymptomatic hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in the study and signed the informed consent.
* Male and female aged between 18 and 65 years old , regardless of gender.
* Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) in the range of (19-30) kg/m2 (including 19 and 30), and no central obesity (waist circumference <90 cm for men, waist circumference <85 cm for women);
* Patients diagnosed as "hyperuricemia" according to The Chinese Guidelines for the Diagnosis and Treatment of Hyperuricemia and Gout (2019), namely, patients whose blood uric acid level exceeds 480 μmol/L twice on other days, and no clinical symptoms related to hyperuricemia such as arthritis;
* Agree to use effective contraceptive methods (including but not limited to abstinence, physical or hormonal contraception, but not hormonal contraception during the study) from signing the informed consent form until 6 months after the infusion of the study drug;
* The subjects can attend the interview on time and complete the interview content.

Exclusion Criteria:

* People who have a history of gout and are using or have used other medications to control uric acid levels in the last 3 months, Asymptomatic hyperuricemia patients who stopped taking uricate-lowering drugs for more than 3 months were excluded.
* Secondary hyperuricemia (such as kidney disease, blood system disease, tumor chemotherapy or drug induced).
* Urolithiasis, or renal, ureteral calculi, urate crystal deposition indicated by ultrasound during screening; The presence of tophi or joint/bursa involvement was indicated by junction ultrasonography.
* Autoimmune disease, allergic disease, prior known food or drug allergy.
* Allergic reactions to recombinant proteins or pig products, or to uricase, polyethylene glycol, corticosteroids and antihistamines.
* Patients who have previously been treated with pegyluricase or other recombinant uricase, or who have been treated with other pegylated biological products.
* Patients have unstable angina, severe arrhythmias requiring drug intervention, congestive heart failure (NYHA grade≥Ⅱ), uncontrolled hypertension (over 150/95 mmHg), poor glycemic control in diabetics ( HbA1c≥7%), end-stage renal disease (CKD4-5), acute stroke, chest imaging suggesting active or severe lung disease, requiring dialysis, organ transplant recipients, and patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Serum creatinine was 1.5 times higher than the upper limit of normal value, and serum transaminase baseline level was 1.5 times higher than the upper limit of normal value.
* Hepatitis B surface antigen positive, hepatitis C antibody positive, treponema pallidum antibody positive or HIV antibody positive in serum virology examination.
* Patients who have been treated with any other investigational drug or participated in another interventional clinical trial within 3 months prior to screening.
* Patients complicated with malignant tumor or undergoing anti-tumor therapy.
* Patients have serious mental and psychological disorders, cognitive disorders and the existence of a history of mental illness.
* Patients have been alcohol abuse within 3 months prior to screening (drinking more than 14 units of alcohol per week (1 unit ≈360 mL beer or 45 mL 40% spirits or 150 mL wine)); Alcohol breath test positive at screening or admission.
* Patients who smoked more than 5 cigarettes a day during the 3 months prior to the study and were unwilling to stop smoking during the study period.
* Patients had been excessive drinking of tea , coffee or caffeinated beverages for a long time (more than 8 cups per day, 1 cup =250 mL); Or any food or beverage containing caffeine or xanthine (such as coffee, strong tea, chocolate, etc.) within 48 hours prior to initial administration.
* Patients have a history of drug or substance abuse, or a positive drug screening test.
* Women who are pregnant or breast-feeding or who plan to become pregnant or breast-feeding during the study period, or who have a positive pregnancy test at the screening stage or baseline.
* The investigator considers that the patient has any other medical or psychological conditions that may pose an undue risk to the subject or interfere with the subject's ability to comply with study protocol requirements or complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
The number of any adverse events (AE) | 35 days after the last dose
  All subjects were observed during the trial for any AE that occurred during the clinical study, including clinical symptoms and life abnormal physical signs, abnormalities in electrocardiogram and laboratory tests. Attention should be paid to the occurrence of AE related to infusion reaction, allergic reaction, vomiting and watery stools/loose stools, acute attack of gout, cardiovascular adverse events and so on.
The number of serious adverse events (SAE) | 35 days after the last dose
  That is serious adverse events, any serious adverse events that occurred to the subject during the study period.

SECONDARY OUTCOMES:
AUC 0-t (Area Under The Plasma Concentration Versus Time Curve) | 35 days after the last dose
  Area under the blood concentration-time curve from 0 to T. It shows the degree to which a drug is absorbed and used in the body.
Cmax(Peak Plasma Concentration) | 35 days after the last dose
  It shows the highest plasma concentration of a drug that can be achieved after administration.
AUC inf (Area Under The Plasma Concentration Versus Time Curve) | 35 days after the last dose
  Area under the blood concentration-time curve from 0 to unlimited time. It shows the degree to which a drug is absorbed and used in the body.
Tmax(Peak Time) | 35 days after the last dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the subject plasma concentration curve after administration.
T ½(Terminal elimination half-life) | 35 days after the last dose
  It reflects how quickly the drug is eliminated from the body.
CL(Clearance Rate) | 35 days after the last dose
  Apparent volume of drug distribution removed from the body per unit time.
The uric acid to creatinine ratio in Urine | 35 days after the last dose
  To evaluate the effect of single use of peruricase on uric acid to creatinine ratio (UAc:Cr) in 24h urine of patients with hyperuricemia.
Vd(Apparent volume of distribution) | 35 days after the last dose
  Apparent volume of distribution refers to the ratio of the amount of drug in vivo to the concentration of drug in blood when a drug reaches dynamic equilibrium in the body. It is a widely used parameters for drug distribution.
λz | 35 days after the last dose
  Elimination rate constant of a drug.It is a common pharmacokinetic indicator.
The positive rate of anti-uricase antibody | 35 days after the last dose
  An evaluation index of immunogenicity of an experimental drug. If detected, it is positive.
The positive rate of anti-PEG antibody | 35 days after the last dose
  An evaluation index of immunogenicity of an experimental drug. If detected, it is positive.
The positive rate of anti-PEG-uricase antibody | 35 days after the last dose
  An evaluation index of immunogenicity of an experimental drug. If detected, it is positive.
Antibody titer of anti-uricase antibody | 35 days after the last dose
  An evaluation index of immunogenicity of an experimental drug.
Antibody titer of anti-PEG Antibody | 35 days after the last dose
  An evaluation index of immunogenicity of an experimental drug.
Antibody titer of anti-PEG-uricase Antibody | 35 days after the last dose
  An evaluation index of immunogenicity of an experimental drug.
Positive rate of neutralizing antibody(NAb) | 35 days after the last dose
  NAb positive rate was assessed by detecting neutralizing antibodies in blood samples.

OTHER OUTCOMES:
pUox(Plasma uricase activity) | 35 days after the last dose
  Plasma uricase activity (pUox) of subjects after single use of peruricase.

CONTACTS AND LOCATIONS:
Overall Officials: The First Affiliated Hospital of Bengbu Medical College The First Affiliated Hospital of Bengbu Medical College, Master, Study Director — Shanghai Institute Of Biological Products; Huan Zhou, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- The first affiliated hospital of Bengbu medical college, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No